CLINICAL TRIAL: NCT07062835
Title: Domestic Perioperative Preparation Application Developed for Children and Parents: Digital Serious Health Game-PeroPap (Perioperative Paediatric Application)
Brief Title: Perioperative Preparation Application Developed for Children and Parents
Acronym: Perioperative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dilek Kucuk Alemdar (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor-Investigator, Dilek Kucuk Alemdar, Professor, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KAEK145; 2023-A4-04-38223 (Other Grant/Funding Number: TÜSEB)
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Surgery
Keywords: children, day surgery , Perioperative, Application

STUDY DESIGN:
Intervention Model Description: The research will be carried out as a prospective, randomised, controlled experimental study.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: After the children who meet the inclusion criteria are randomly assigned to the study groups, the children and their parents will be informed which group they are included in and their written consent will be obtained through the informed consent form. Since the project coordinator will provide information about the use of the application, it will not be blinded. However, the doctor who will perform the surgery will not know which group the children are in. In addition, in order to prevent detection bias, the output measurements of the study will be made by the nurse who does not know who is in the experimental group and who is in the control group. In order to prevent bias in the evaluation of the data, the study groups will be coded in the database as A and B by a person outside the scope of the research, and the data will be analyzed by a statistical expert independent of the research. It was aimed to prevent statistical and reporting bias by blinding in terms of output measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative Paediatric Application Group (Experimental): Children in the experimental group will start receiving interactive perioperative preparation training with the PeroPap application 1 day before surgery and play the PeroPap game. Children will learn about the operation process by watching and playing the PeroPap character's cartoon story about the operation process. They will also listen to the song "PeroPap is having surgery" and play the "PeroPap Game" in the application, which they can play before and after surgery.
  Interventions: Behavioral: Perioperative Paediatric Application
- Control (Active Comparator): . In order to meet the perioperative health care needs of the children and their parents in the control group, when they applied to the outpatient clinic for anaesthesia consultation on the working day before the operation, standard individualised care interventions will be provided according to their needs preoperatively and until their discharge, and children and parents will be given surgery preparation training with the education booklet "PeroPap is Having Surgery".
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Perioperative Paediatric Application — Children in the experimental group will start receiving interactive perioperative preparation training with the PeroPap application 1 day before surgery and play the PeroPap game. Children will learn about the operation process by watching and playing the PeroPap character's cartoon story about the operation process. They will also listen to the song "PeroPap is having surgery" and play the "PeroPap Game" in the application, which they can play before and after surgery. At the same time, in the parent module, information will be provided for parents with the cartoon story "PeroPap is Having Surgery".
  Arms: Perioperative Paediatric Application Group
Other: Control — In order to meet the perioperative health care needs of the children and their parents in the control group, when they applied to the outpatient clinic for anaesthesia consultation on the working day before the operation, standard individualised care interventions will be provided according to their needs preoperatively and until their discharge, and children and parents will be given surgery preparation training with the education booklet "PeroPap is Having Surgery".
  Arms: Control

SUMMARY:
Approaches to increase the compliance of children and parents in daily surgical interventions in children are limited. The primary aim of this study is to evaluate the clinical usability of the Paediatric Perioperative Preparation Game Application-PeroPap, which will be developed to prepare children and parents for day surgery. The secondary aim is to investigate its effect on the perioperative adaptation process of children and parents, children's symptoms such as pain, anxiety, nausea, vomiting and postoperative behavioural changes, and parents' anxiety and satisfaction.

DETAILED DESCRIPTION:
Approaches to increase the compliance of children and parents in daily surgical interventions in children are limited. The primary aim of this study is to evaluate the clinical usability of the Paediatric Perioperative Preparation Game Application-PeroPap, which will be developed to prepare children and parents for day surgery. The secondary aim is to investigate its effect on the perioperative adaptation process of children and parents, children's symptoms such as pain, anxiety, nausea, vomiting and postoperative behavioural changes, and parents' anxiety and satisfaction. The research will be carried out as a prospective, randomised, controlled experimental study in the Pediatric Surgery Clinic of Ordu University Training and Research Hospital Gynecology and Children's Hospital. The population of the study will consist of children aged 7-10 years who underwent day surgery between the dates of the study. The sample of the study will consist of 348 children and their parents who will undergo day surgery between the specified dates, who meet the case selection criteria and agree to participate in the study. The study participants will be assigned to two groups as experimental (n=174) and control group (n=174) by computer-assisted randomisation. In the first phase of the study, PeroPap design will be created with expert opinions using the serious game development framework. The digital serious health game application PeroPap will be developed as an evidence-based interactive game specifically designed to address relevant challenges faced by the user and change behaviour. Children and parents will be downloaded to their digital devices with Android or IOS operating system by scanning the QR code by the executive via internet connection. Two separate options will be created for the child and parent on the application. Children in the experimental group will start receiving interactive perioperative preparation training with the PeroPap application 1 day before surgery and play the PeroPap game. Children will learn about the operation process by watching and playing the PeroPap character's cartoon story about the operation process. They will also listen to the song "PeroPap is having surgery" and play the "PeroPap Game" in the application, which they can play before and after surgery. At the same time, in the parent module, information will be provided for parents with the cartoon story "PeroPap is Having Surgery". The application will also include deep breathing exercises and mindfulness practices to reduce parents' anxiety. In order to meet the perioperative health care needs of the children and their parents in the control group, when they applied to the outpatient clinic for anaesthesia consultation on the working day before the operation, standard individualised care interventions will be provided according to their needs preoperatively and until their discharge, and children and parents will be given surgery preparation training with the education booklet "PeroPap is Having Surgery". Research data will be collected with the Child and Parent Descriptive Information Form, Child Perioperative Follow-up Form, Baxter Nausea Scale-BARF, Eastern Ontario Children's Hospital Pain Scale, Comfort Behaviours Checklist (CBCL), Multidimensional Perioperative Anxiety Scale in Children, Modified Yale Preoperative Anxiety Scale, Postoperative Pain Scale for Parents, State and Trait Anxiety Scale and PedsQL Health Care Parent Satisfaction Scale.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 7 and 10 years old,
* The child receives general anesthesia
* The child is hospitalized for a surgical operation,
* Voluntariness of parents and children to participate in the study,
* The child has no visual, hearing or mental disabilities,
* The parent or child has an Android or IOS device with an internet connection,
* Written and verbal consent from parents and children.

Exclusion Criteria:

* The child has a hearing problem,
* The child and parent are not comfortable speaking and understanding Turkish,
* The child is not at the level of mental development to answer the questions asked,
* Lack of a primary caregiver.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale: | 1 day before surgery, 1 hour before surgery, 15 minutes before surgery, 1 hour and 2 hours after surgery.
  In this scale, there are 22 items under 5 categories (activity, speech, emotional state, degree of arousal, relationship with family), each representing a different area of the child's anxiety, and the pediatric patient is evaluated at different points in the preoperative phase. Each category is calculated by taking a score between 0 and 4 (0-6 for the speech category) according to the patient's behavior. During the calculation, a total score of 33-100 is obtained by multiplying the decimal values obtained by dividing the score between 0-4 divided by 4 for 4 categories consisting of 4 items by the decimal value obtained by dividing the score between 0-6 divided by 6 for 1 category consisting of 6 items by 20 (100/total number of categories)
Eastern Ontario Children's Hospital Pain Scale | Postoperative 1st hour and 2nd hour.
  The scale evaluates six sub-items of the scale including crying, facial expression, verbal expression, body, touch, and legs in the postoperative period. In the scale; the first item (Crying) can score a minimum of 1 point and a maximum of 3 points, items 2 (Facial expression) and 3 (Verbal expression) can score a minimum of 0 points and a maximum of 2 points, items 4 (Body), 5 (Touch) and 6 (Legs) can score a minimum of 1 point and a maximum of 2 points. The total score from the scale is evaluated as a minimum of 4 and a maximum of 13 points. A high total score on the scale indicates that the child has high pain in the postoperative period.
Multidimensional Perioperative Anxiety Scale: | 1 day before surgery, 1 hour before, 15 minutes before, 1 hour and 2 hours after surgery.
  The scale is a visual analog scale prepared for children between the ages of 7-13 who will undergo day surgery, consisting of 5 items and scored between 0-100. An increase in the score obtained from the scale indicates that the child's perioperative anxiety increases
Comfort Behavior Checklist (CBCL): | 1 hour and 2 hours after surgery.
  The PACCL consists of 30 behavioral indicators, pain and comfort scores. High scores indicate a high comfort level. If all questions are answered, the minimum score that can be obtained from the scale is 25 and the maximum score is 100

SECONDARY OUTCOMES:
PedsQL Health Care Parental Satisfaction Scale | 30 minutes before discharge
  The questions in the scale aim to measure satisfaction with health care services and psychosocial satisfaction. The scale consists of 25 questions with 6 subheadings: information, family involvement, communication, technical skills, emotional needs and general satisfaction. The questions in the scale are evaluated on a 5-point scale. "0" means never satisfied, "1" means sometimes satisfied, "2" means most of the time satisfied, '3' means almost always satisfied, "4" means always satisfied.
Postoperative Pain Scale for Parents: | 1 hour and 2 hours after surgery.
  It allows parents to assess pain at different times of the day for postoperative pain measurement. The scale includes 15 items, each with a "Yes" or "No" response. Questions with a "Yes" answer are scored and the total score that can be obtained from the scale is at least 15. Scores between 6 and 15 on the scale indicate that "the child has clinically significant pain", while a score between 0 and 6 on the EPAS indicates that the child has pain that does not require intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Altinordu, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No